CLINICAL TRIAL: NCT04179357
Title: Hemostatic Disorders Impact on Intensive Care Patients.
Brief Title: Hemostatic Disorders on Intensive Care Patients.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Fawzi Ibrahim Mansour, Resident Doctor, Assiut University
Other Study IDs: Hemostatic Disorders
Record Dates: First submitted 2019-09-24; First posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Hemostatic Disorder
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To assess the incidence of hemostatic disorders among ICU patients.
2. To establish a relationship between supportive treatment and survival in patients with coagulopathy in ICU.
3. To provide solutions that can help in reduction of the incidence of hemostatic disorders in ICU patients.

DETAILED DESCRIPTION:
Hemostasis is the physiological process that stops bleeding at the site of an injury while maintaining normal blood flow elsewhere in the circulation. Blood loss is stopped by formation of a hemostatic plug. The endothelium in blood vessels maintains an anticoagulant surface that serves to maintain blood in its fluid state, but if the blood vessel is damaged components of the subendothelial matrix are exposed to the blood. Several of these components activate the two main processes of hemostasis to initiate formation of a blood clot, composed primarily of platelets and fibrin.

Many critically ill patients develop hemostatic abnormalities, ranging from isolated thrombocytopenia to complex defects, such as DIC. Coagulation abnormalities are commonly found in critically ill patients. Prompt and proper identification of the underlying cause of these coagulation abnormalities is required, since each coagulation disorder necessitates very different therapeutic management strategies.

Management of coagulopathy The key basic management principle of all coagulopathies is that the decision to transfuse blood products should not be based on the results of coagulation tests alone, rather an individualized approach is warranted. It is imperative to synthesizes all the available clinical data and treat the underlying cause.

In summary, hemostatic disorders are very common in the critically ill. Blood product support is frequently required, but there is only a very limited evidence-base to support its use. In many cases, no specific product support is required and the key management step is the treatment of the condition underlying the coagulopathy .

ELIGIBILITY:
Inclusion Criteria:

* Intensive care unit patients,aged more than 18 years .
* Any Acquired bleeding disorders (platelet disorders; thrombocytopenia, acquired thrombocythemia and thrombocytosis, acquired coagulation defect, Thrombophilia ) Diagnosed in Critical care unit in Assiut university in one year time frame

Exclusion Criteria:

* Patient less than 18 years.
* Patients with Inherited platelet defects ( Amegakaryoctye aplasia and Bernard Soulir syndrome)
* Patients with Inherited coagulation defects (e.g.hemophilia , Von Willebrand disease and any inherited coagulation defect.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All cases who will be admitted at the intensive care units at Assiut university Hospital through 1 year duration .
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Describe the Pattern of Homeostasis Disorders occur in Critical Care Unit in Assiut University | Baseline
  Study the causes of either bleeding or thrombotic events in Critical care unit. Describe the pattern of the disease regarding age, sex and predisposing factors.

SECONDARY OUTCOMES:
Correlate Supportive and Definitive Treatment and Outcomes of Patients with Homeostasis Disorder in ICU. | Baseline
  Study the forms of transfusion ( e.g.packed red blood cells, Platelet , Fresh frozen plasma), anti bleeding measures (e.g. Tranexamic acid), anticoagulant and anti platelet drugs received by the patients and their outcomes

REFERENCES:
- [Background] Retter A, Barrett NA. The management of abnormal haemostasis in the ICU. Anaesthesia. 2015 Jan;70 Suppl 1:121-7, e40-1. doi: 10.1111/anae.12908. PMID 25440406
- [Background] Hunt BJ. Bleeding and coagulopathies in critical care. N Engl J Med. 2014 Feb 27;370(9):847-59. doi: 10.1056/NEJMra1208626. No abstract available. PMID 24571757